CLINICAL TRIAL: NCT03855696
Title: A Phase I, Randomized, Double-blind, Placebo-Controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MG1113 in Healthy Subjects and Hemophilia Patients
Brief Title: A Study to Investigate the Safety, Tolerability, PK and PD of MG1113 in Healthy Subjects and Hemophilia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Dream CIS, Inc. (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: MG1113_P1
Record Dates: First submitted 2019-02-12; First posted 2019-02-27 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia
Keywords: MG1113; Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation model
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MG1113 (Experimental): * Anti-tissue factor pathway inhibitor (TFPI) recombinant antibody
  * Each vial contains 1mL of study drug
  * The doses planned in healthy subjects are 0.5 mg/kg, 1.7 mg/kg, and 3.3 mg/kg by SC injection; 3.3 mg/kg by IV injection. In hemophilia patients, 1.7 mg/kg and 3.3 mg/kg will be administered by SC injection.
  Interventions: Biological: MG1113
- Placebo of MG1113 (Placebo Comparator): * Placebo of MG1113
  * Each vial contains 1mL of study drug
  Interventions: Other: Placebo of MG1113

INTERVENTIONS:
Biological: MG1113 — MG1113
  Arms: MG1113
Other: Placebo of MG1113 — Placebo of MG1113
  Arms: Placebo of MG1113

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MG1113 in the single ascending dose study (IV injection or SC injection) in healthy subjects and hemophiia patients.

DETAILED DESCRIPTION:
This is a single-dose study that explore the safety, tolerability, PK, and PD of the study drug by sequentially increasing the study drug in 4 dose levels. The route of administration is either subcutaneous (SC) injection or intravenous (IV) injection.

For healthy subjects, 6 subjects will be assigned to the study group and 2 subjects will be assigned to the placebo group to explore the safety and tolerability, and PK/PD of the study drug in comparison with placebo. Hemophilia patients will be assigned only to the study group with 3 and 6 subjects in each cohort, respectively.

The investigator and subjects will know which cohort the healthy subjects have been assigned to, but they will be double-blinded as to whether the subjects are assigned to the study group (study drug) or the placebo group (placebo) within each cohort.

The doses planned in healthy subjects are 0.5 mg/kg, 1.7 mg/kg, and 3.3 mg/kg by SC injection; 3.3 mg/kg by IV injection. In hemophilia patients, 1.7 mg/kg and 3.3 mg/kg will be administered by SC injection. The planned dose will be administered after checking the safety and tolerability at the previous dose to the extent not exceeding the criteria for discontinuation of dose escalation. The dose escalation will be decided by the Data Monitoring Committee(DMC) and Data and Safety Monitoring Boards (DSMB) in the blinded evaluation of the safety and tolerability data obtained from each previous cohort for 7 days after administration. Before deciding dose escalation and proceeding to the next step, the safety, tolerability, PK, and PD data obtained from all healty subjects and hemophilia patients up to cohort 6 will be evaluated by the Data and Safety Monitoring Boards (DSMB) in an unblinded manner. In addition, if necessary, the analysis result of cohort that has completed all the scheduled visits can be reviewed in an unblinded manner.

ELIGIBILITY:
<Healthy adult subjects>

* Inclusion Criteria:

  1. Healthy male adult subjects aged 19-60 years (both inclusive) at screening
  2. 50 to 90 kg in weight with calculated BMI between 18.5 and 29.9 kg/m2
  3. Agree to use medically acceptable adequate dual contraceptive methods (condom, vasectomy, spermicide, oral contraceptives, intrauterine device, and complete sexual abstinence, etc.) and not to donate sperm until 3 months after administration of the investigational product
  4. Voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a detailed explanation on this study and fully understanding the information
* Exclusion Criteria:

  1. Presence or history of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immune, skin, nervous, or psychiatric disease
  2. Symptoms of acute disease within 28 days of investigational product administration
  3. Medical history that may affect absorption, distribution, metabolism and excretion of drugs
  4. Clinically significant active chronic disease
  5. Clinically significant allergic disease (however, mild allergic rhinitis or allergic dermatitis not requiring any medication is allowed) or history of any anaphylactic reaction
  6. Any of the following results from laboratory tests: 1) AST (sGOT) or ALT (sGPT) >2 x UNL 2) Hb < 9.0 g/dL 3) Absolute Neutrophil Count < 1500 mm2 4) Platelet count < 100 x 103 mm2 5) aPTT, PT > 1.5 x UNL 6) Have hepatitis B (HBsAg positive) or C (anti-HCV positive), or have positive HIV test result 7) Creatinine clearance ≤80 mL/min (calculated by the Cockcroft-Gault formula)
  7. Have a family history or be considered to be at risk of thromboembolic events, or have the following test results: 1) Antithrombin level ≤LNL 2) Protein C or S activity ≤LNL 3) Factor V Leiden mutation 4) Prothrombin G20210A mutation
  8. Used ethical drugs including prescription drugs within 14 days of investigational product administration
  9. Used drugs (over-the-counter drugs, herbal medicines, and nutritional agents and vitamins for the purpose of same efficacy) within 7 days of investigational product administration
  10. Cannot have standard meals provided at the hospital
  11. Donated whole blood within 60 days of investigational product administration, or donated blood components within 20 days of investigational product administration, or received blood transfusion within 1 month before administration
  12. Participated in another clinical trial or bioequivalence study within 90 days of investigational product administration (If participating in a clinical trial after 12/06/2019, not within 90 days, but within 6 months is applied)
  13. Individuals who consume caffeine (caffeine >5 cups/day) or alcohol (alcohol >30 g/day) continuously, who cannot abstain from drinking during the study, or heavy smoker (>10 cigarettes/day)
  14. Determined to be ineligible to participate in the study per investigator's judgment due to other reasons including the laboratory test results
  15. History of drug abuse or positive urine drug screen results

<Hemophilia patients>

* Inclusion criteria

  1. Male hemophilia A or B patients aged 19-60 years (both inclusive) at screening
  2. ≥50 kg in weight with calculated BMI between 18.5 and 29.9 kg/m2
  3. Agree to use medically acceptable adequate dual contraceptive methods (condom, vasectomy, spermicide, oral contraceptives, intrauterine device, and complete sexual abstinence, etc.) and not to donate sperm until 60 days after administration of the investigational product
  4. Voluntarily decided to participate in the study and provided written consent to follow precautions after receiving a detailed explanation on this study and fully understanding the information
* Exclusion criteria

  1. Symptoms of acute disease within 28 days of investigational product administration or any surgery planned during the study period
  2. Medical history that may affect absorption, distribution, metabolism and excretion of drugs
  3. Clinically significant active chronic disease
  4. Clinically significant allergic disease (however, mild allergic rhinitis or allergic dermatitis not requiring any medication is allowed) or history of any anaphylactic reaction
  5. Patients having current human factor VIII or IX with an inhibitor titer of >5 Bethesda units or patients requiring treatment with bypassing agent
  6. Patients who has a history of confirmed human factor VIII or IX with an inhibitor titer of >5 Bethesda units at any time
  7. History of ≥6 bleeding episodes despite temporary bypassing agent administered for 24 weeks before screening, or ≥2 bleeding episodes despite the bypassing agent administered prophylactically
  8. Received factor VIII or factor IX within 48 hours prior to administration of the investigational product
  9. Hemostatic agent, etc. prescribed to control bleeding within 5 days prior to administration of the investigational product
  10. Immune tolerance induction prescribed within 30 days prior to administration of the investigational product
  11. Currently using systemic immunomodulator (e.g., interferon or rituximab)
  12. Be at risk of thrombotic microangiopathy per investigator's judgment or have related medical history or family history
  13. Congenital or acquired anticoagulant disorders other than hemophilia A or B, or conditions of other diseases that increase the risk of bleeding or thrombus (e.g., autoimmune disease)
  14. Any of the following results from laboratory tests: 1) AST (sGOT) or ALT (sGPT) >3 x UNL 2) Hb < 9.0 g/dL 3) Absolute Neutrophil Count < 1500 mm2 4) Platelet count < 100 x 103 mm2 5) Have hepatitis B (HBs Ag positive) or C (anti-HCV positive), or have HIV positive test result 6) Creatinine clearance ≤80 mL/min (calculated by the Cockcroft-Gault formula)
  15. Cannot have standard meals provided at the hospital
  16. Participated in another clinical trial within 90 days of investigational product administration
  17. Individuals who consume caffeine (caffeine >5 cups/day) or alcohol (alcohol >30 g/day) continuously, who cannot abstain from drinking during the study, or heavy smoker (>10 cigarettes/day)
  18. Determined to be ineligible to participate in the study per investigator's judgment due to other reasons including the laboratory test results
  19. History of drug abuse or positive urine drug screen results

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | Through study completion (~50 day)
  Adverse events such as subjective and objective symptoms

SECONDARY OUTCOMES:
Immunogenicity assay | Through study completion (~50 day)
  ADA [Anti-Drug Ab]
Pharmacokinetic assessment - Cmax | Through study completion (~50 day)
  Cmax
Pharmacokinetic assessment - Tmax | Through study completion (~50 day)
  Tmax
Pharmacokinetic assessment - AUClast | Through study completion (~50 day)
  AUClast
Pharmacokinetic assessment - AUCinf | Through study completion (~50 day)
  AUCinf
Pharmacokinetic assessment - half-life | Through study completion (~50 day)
  half-life
Pharmacokinetic assessment - CL/F (for SC) | Through study completion (~50 day)
  CL/F (for SC)
Pharmacokinetic assessment - CL (for IV) | Through study completion (~50 day)
  CL (for IV)
Pharmacokinetic assessment - Vd/F (for SC) | Through study completion (~50 day)
  Vd/F (for SC)
Pharmacokinetic assessment - Vd (for IV) | Through study completion (~50 day)
  Vd (for IV)
Pharmacokinetic assessment - Bioavailability (F) | Through study completion (~50 day)
  Bioavailability (F) Bioavailability (F) = AUCinf (at SC dosing [3.3 mg/kg])/AUCinf (at IV dosing [3.3 mg/kg])
Pharmacodynamic assessment - Free TFPI in plasma | Through study completion (~50 day)
  Free TFPI in plasma (ng/mL)
Pharmacodynamic assessment - Diluted PT | Through study completion (~50 day)
  Diluted PT (sec)
Pharmacodynamic assessment - residual TFPI activity | Through study completion (~50 day)
  residual TFPI activity
Pharmacodynamic assessment - Thrombin generation | Through study completion (~50 day)
  Thrombin generation (lag time, peak generation, Endogenous thrombin generation potential [ETP])
Pharmacodynamic assessment - Pro-coagulant effect | Through study completion (~50 day)
  Pro-coagulant effect (D-dimer, Fibrinogen, prothrombin fragments 1+2)
Physical examination | Through study completion (~50 day)
  Physical examination
Incidence of participant abnormalities in 12-lead ECG (Ventricular rate in beat/min, Interval for PR in msec, QRS in msec, QTc in msec) for physiological parameter | Through study completion (~50 day)
  The result for 12-lead ECG will be reported as Clinical Significant or Not-Clinical Significant.
  * Ventricular rate in beat/min
  * Interval for PR in msec
  * QRS in msec
  * QTc in msec
Vital signs - blood pressure (Systolic, Diastolic) | Through study completion (~50 day)
  Vital signs - blood pressure (Systolic, Diastolic)
Vital signs - pulse rate | Through study completion (~50 day)
  Vital signs - pulse rate
Vital signs - body temperature | Through study completion (~50 day)
  Vital signs - body temperature
Frequency of Bleeding (only for hemophilia patients) | Through study completion (~50 day)
  Bleeding evaluation (only for hemophilia patients) by questionnaire; Occurrence date, Persistence in yes or no questionnaire, Causes (blood in naturally occurring/Traumatic bleeding), Severity (mild/moderate/Severe)
Local reaction in injection site | Through study completion (~50 day)
  Pain or tenderness, itching, rash, redness (in mm), and induration (in mm) will be reported.
  Local stimulation test in injection site: Occurrence date, Persistence, Causes, Severity (mild/moderate/Severe) The occurrence of pain or tenderness, itching and rash will be reported by Yes or No questionnaire.
  The size of redness and induration will be measured in millmeters(mm).
Incidence of participant abnormalities in laboratory tests by physiological parameter (Hematology, clinical chemistry, urinalysis, and blood coagulation test) | Through study completion (~50 day)
  Parameters for laboratory tests include Hematology(WBC in 10**3/mcL,Neutrophils in %,ANC in mcL,Lymphosyte in %,Monocyte in %,Eosinophils in %,Basophils in %,RBC in 10**6/mcL,Hemoglobin in g/dL,Hematocrit in %,MCV in fL, MCH in pg,MCHC in g/dL,Platelets in 10**3/mcL,MPV in fL),Clinical chemistry(Glucose in mg/dL,BUN in mg/dL,Uric adic in mg/dL,Total cholesterol in mg/dL,Triglyceride in mg/dL,Protein,Albumin in g/dL,Total bilirubin in mg/dL,Alkaline phosphatase in IU/L,AST in IU/L,ALT in IU/L,r-GT in IU/L,LDH in IU/L,Serum creatinine in mg/dL,Na in mmol/L,K in mmol/L,Cl in mmol/L,CPK in IU/L,Troponin I in ng/mL,Troponin T in ng/mL,Creatinine Clearance),Urinalysis(These values are reported only as a number;Specific garavity,Color,pH,Protein,Glucose,Ketone,Bilirubin,Blood,Urobilinogen,Nitrite,WBC,Squma EP cell,Casts,Crystal,Clarity,RBC),Blood coagulation test (aPTT in sec,PT in sec,Fibronogen in mg/dL,Antithrombon III in %,Protein C in %,Protein S in%)

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, MD, Principal Investigator — Korea University Anam Hospital
Locations (2):
- South Korea (2):
  - Yonsei Cancer Center, Yonsei University Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No